CLINICAL TRIAL: NCT04828681
Title: Functional Coronary Angiography-Derived Index of Microcirculatory Resistance and Microvascular Obstruction in Cardiac Magnetic Resonance Imaging After ST-segment Elevation Myocardial Infarction
Brief Title: Angio-IMR and Cardiac MR-derived MVO in STEMI Patients
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Collaborators: RainMed Medical Group (Industry); Shanghai Institute of Cardiovascular Diseases (Other)
Responsible Party: Principal Investigator, Joo Myung Lee, Assistant Professor, Samsung Medical Center
Other Study IDs: SMCCMR88848439
Record Dates: First submitted 2021-03-30; First posted 2021-04-02 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: ST-segment Elevation Myocardial Infarction (STEMI)
Keywords: ST-segment Elevation Myocardial Infarction (STEMI); Index of microcirculatory resistance; Cardiac magnetic resonance imaging; Microvascular obstruction; Coronary microcirculation
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Angio-IMR>40 Unit: Patients with angio-IMR>40U in the culprit vessel after successful primary PCI.
  Interventions: Diagnostic Test: Cardiac magnetic resonance imaging
- Patients with Angio-IMR≤40 Unit: Patients with angio-IMR≤40U in the culprit vessel after successful primary PCI.
  Interventions: Diagnostic Test: Cardiac magnetic resonance imaging

INTERVENTIONS:
Diagnostic Test: Cardiac magnetic resonance imaging — Cardiac magnetic resonance imaging was performed 5.0 ± 5.8 days after the primary PCI. MVO, infarct size, and myocardial salvage index were quantitatively assessed in CMR.

SUMMARY:
Coronary microcirculatory dysfunction has been known to be prevalent even after successful revascularization of ST-segment elevation myocardial infarction (STEMI) patients. Microvascular obstruction (MVO) in cardiac magnetic resonance (CMR) is significant prognostic indicator in STEMI patients after primary percutaneous coronary intervention (PCI). Although current gold-standard method to assess microvascular damage or dysfunction in STEMI patients is CMR and assessment of MVO, previous study presented that index of microcirculatory resistance (IMR) in culprit vessel of STEMI patients showed significant association with the presence of MVO in CMR and the risk of cardiac death or heart failure admission. Nevertheless, the need for pressure-temperature sensor wire and hyperemic agents significantly limits adoption of IMR in daily practice.

Recent technical development enabled angiographic derivation of IMR without pressure wire, hyperemic agents, or thermodilution method. In this regard, the current study will evaluate the feasibility of functional angiography-derived IMR (angio-IMR) in the evaluation of MVO after successful primary PCI for STEMI.

DETAILED DESCRIPTION:
Coronary microcirculatory dysfunction has been known to be prevalent even after successful revascularization of ST-segment elevation myocardial infarction (STEMI) patients. Microvascular obstruction (MVO) in cardiac magnetic resonance (CMR) is significant prognostic indicator in STEMI patients after primary percutaneous coronary intervention (PCI). Although current gold-standard method to assess microvascular damage or dysfunction in STEMI patients is CMR and assessment of MVO, previous study presented that index of microcirculatory resistance (IMR) in culprit vessel of STEMI patients showed significant association with the presence of MVO in CMR and the risk of cardiac death or heart failure admission. Nevertheless, the need for pressure-temperature sensor wire and hyperemic agents significantly limits adoption of IMR in daily practice.

Recent technical development enabled angiographic derivation of IMR without pressure wire, hyperemic agents, or thermodilution method. In this regard, the current study will evaluate the feasibility of functional angiography-derived IMR (angio-IMR) in the evaluation of MVO after successful primary PCI for STEMI.

The study population will be derived from the prospective institutional AMI registry of Samsung Medical Center between December 2007 and July 2014. Main results from this registry were published elsewhere (PLoS One. 2017 Jan 12;12(1):e0170115 and Sci Rep. 2019 Jul 4;9(1):9646). In this registry, 515 consecutive patients who presented with acute myocardial infarction and underwent CMR were prospectively enrolled. AMI was defined as evidence of myocardial injury (defined as elevation of cardiac troponin values, with at least one value above the 99th percentile upper reference limit) with necrosis in a clinical setting, consistent with myocardial ischemia. Among the total patients, STEMI patients (n = 332), whose electrocardiogram showed ST-segment elevation more than 1 mm in two or more contiguous leads or a presumably new-onset left bundle branch block, will be analyzed for the current study. For the study purpose, patients with failed primary PCI (n=1), treated by medical treatment alone without PCI (n=4), and no available coronary angiographic images (n=3) will be excluded. Among the remaining 324 patients, functional coronary angiography core laboratory (Shanghai Institute of Cardiovascular Diseases, Shanghai, China) evaluated the quality of angiographic images and additionally exclude patients with insufficient image quality for angio-IMR calculation (n=37). All patients also underwent baseline and 1-year follow-up echocardiography. The Institutional Review Board of Samsung Medical Center approved this study, and all patients provided written informed consent.

The association of Angio-IMR with CMR-derived quantitative parameters (extent of MVO, infarct size, area at risk) and qualitative parameter (presence of MVO) will be analyzed. The discrimination ability of angio-IMR to predict the presence of MVO in CMR will be compared with conventional angiographic measures of culprit vessel reperfusion (TIMI flow grade, myocardial blush grade).

ELIGIBILITY:
Inclusion Criteria:

* STEMI patients
* Successful primary PCI in the culprit vessel
* Underwent cardiac MR during index hospitalization
* Suitable coronary angiographic images for angio-IMR analysis

Exclusion Criteria:

* patients with failed primary PCI
* treated by medical treatment alone without PCI
* no available coronary angiographic images
* insufficient image quality for angio-IMR calculation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be derived from the prospective institutional AMI registry of Samsung Medical Center between December 2007 and July 2014. In this registry, 515 consecutive patients who presented with acute myocardial infarction and underwent CMR were prospectively enrolled. Among the total patients, STEMI patients (n = 332) will be analyzed for the current study. For the study purpose, patients with failed primary PCI (n=1), treated by medical treatment alone without PCI (n=4), and no available coronary angiographic images (n=3) will be excluded. Among the remaining 324 patients, patients with insufficient image quality for angio-IMR calculation will be additionally excluded (n=37).
Sampling Method: Non-Probability Sample
Enrollment: 324 (Actual)
Dates: Start 2007-12-24 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of microvascular obstruction in CMR | At the time of index hospitalization
  Proportion of microvascular obstruction in CMR

SECONDARY OUTCOMES:
Correlation of angio-IMR with the extent of microvascular obstruction in CMR | At the time of index hospitalization
  Correlation of angio-IMR with the extent of microvascular obstruction (% of left ventricular mass) in CMR
Correlation of angio-IMR with the infarct size in CMR | At the time of index hospitalization
  Correlation of angio-IMR with the infarct size (% of left ventricular mass) in CMR
Correlation of angio-IMR with the area at risk in CMR | At the time of index hospitalization
  Correlation of angio-IMR with the area at risk (% of left ventricular mass) in CMR
Correlation of angio-IMR with the myocardial salvage index in CMR | At the time of index hospitalization
  Correlation of angio-IMR with the myocardial salvage index in CMR
Discrimination ability of angio-IMR to predict the occurrence of microvascular obstruction in CMR | At the time of index hospitalization
  area under curve in ROC analysis of angio-IMR to predict the occurrence of microvascular obstruction in CMR
Left ventricular ejection fraction | At the time of index hospitalization and 1 year follow-up
  Left ventricular ejection fraction in echocardiography
Regional wall motion score index | At the time of index hospitalization and 1 year follow-up
  Regional wall motion score index in echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Joo Myung Lee, MD, MPH, PhD, Principal Investigator — Samsung Medical Center
Locations (2):
- University of Iowa Carver College of Medicine, Iowa City, IA, USA, Iowa City, Iowa, United States
- Shanghai Institute of Cardiovascular Diseases, Shanghai, China, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be able to be shared upon reasonable request after discussion by steering committee members and principal investigator.

REFERENCES:
- [Derived] Shin D, Kim J, Choi KH, Dai N, Li Y, Lee SH, Joh HS, Kim HK, Kim SM, Ha SJ, Jang MJ, Park TK, Yang JH, Song YB, Hahn JY, Choi SH, Choe YH, Gwon HC, Lee JM. Functional angiography-derived index of microcirculatory resistance validated with microvascular obstruction in cardiac magnetic resonance after STEMI. Rev Esp Cardiol (Engl Ed). 2022 Oct;75(10):786-796. doi: 10.1016/j.rec.2022.01.004. Epub 2022 Mar 3. English, Spanish. PMID 35249841